CLINICAL TRIAL: NCT03426930
Title: Contribution of a Virtual Reality Program in the Treatment of Dysmorphophobia for Adolescent Female With Anorexia Nervosa
Acronym: TERV-TCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-40; 2017-A02836-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The reference treatment of dysmorphophobia used (Active Comparator)
  Interventions: Other: self-evaluation of the Body Mass Index; Other: Cognitive-behavioral psychotherapies
- The reference treatment with the virtual reality (Experimental)
  Interventions: Other: self-evaluation of the Body Mass Index; Other: Cognitive-behavioral psychotherapies

INTERVENTIONS:
Other: self-evaluation of the Body Mass Index — Evaluation of the Body Mass Index before and after the treatment
Other: Cognitive-behavioral psychotherapies — Cognitive-behavioral psychotherapies before and after the treatment

SUMMARY:
Anorexia nervosa is an eating disorder that begins frequently in adolescence between the ages of 13 and 19, which affects girls with a sex ratio of 10:1, and the prevalence for females varies from 0,3% to 0,9%.

The current therapeutic arsenal has a limited success in the treatment of anorexia nervosa with a long-term mortality rate and a 12-month relapse rate of up to 10% and 40%, respectively.

One of the most difficult symptoms to treat is a body dysmorphic disorder, also called dysmorphophobia, the persistence of this symptom is a major negative prognostic factor.

The main treatment of dysmorphophobia is currently cognitive behavioral therapy (CBT). In most protocols, the technique of progressive exposure face to the mirror is used with low efficiency. Adapted physical activity has recently been proposed in the literature as a tool to improve body perception.

Face of complex management of this major symptom that is dysmorphophobia, some offer to use virtual reality.

It is in this context that the study proposes to study the contribution of virtual reality in the treatment of the body dysmorphic disorder of adolescent patients hospitalized for anorexia nervosa in the department of Child and Adolescent Psychiatry Salvator Hospital in Marseille.

It will be compare the importance and the evolution of the dysmorphophobia between two groups of teenagers hospitalized in Space Arthur for anorexia nervosa: an experimental group receiving the treatment with the contribution of the virtual reality, and a control group receiving the reference treatment of dysmorphophobia used in our unit.

It will be recruit 30 adolescent females with anorexia nervosa according to the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM)-5. The subjects will be divided into 2 groups of 15 teenagers, according to a randomization list, a group with a classic protocol, a group with virtual reality. The subjects with virtual reality will have 5 exposure sessions where they will be able to model their body in view in 1st person and 3rd person, via an Oculus Rift. It will be compare the following parameters: the different scores related to dysmorphophobia according to different questionnaires, the self-evaluation of the Body Mass Index (BMI), in order to observe the evolution of the symptom, then the anxiety relative to the exposure of a BMI higher in order to work the fear of getting fat, the choice of the most pleasant BMI, to evaluate skinny body addiction.

At the end of the study, we hope to highlight the effectiveness of virtual reality to fight against dysmorphophobia, in order to have a better estimate of its body aspect, and to impact the evolution towards the cure in anorexia nervosa in teenage girls. In addition to increasing our knowledge, this could allow to consider new strategies in the management of anorexia nervosa, and why not democratize more virtual reality with adolescents followed in child and adolescent psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 et 18 years old
* Female subject
* Females with anorexia nervosa according to the diagnostic criteria of DSM-5
* The patient, the parents or the legal representative (s) have given written consent
* Possessing a social security scheme

Exclusion Criteria:

* Male subject
* Age under 13 years or over 18 years
* Subject presenting a contra-indication to virtual reality
* Subject, or parents who refused to sign informed consent

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-01-17 (Estimated); Study Completion 2021-01-17 (Estimated)

PRIMARY OUTCOMES:
Evaluation of non-self Body Mass Index | 24 months
  the self-evaluation of BMI will allow to observe the evolution of the symptom of dysmorphophobia. Explicit and implicit assessment of lean body addiction.
Eating Disorder Inventory 2 (EDI) | 24 months
  The EDI is intended to assess attitudes and behaviors related to eating behavior in 11 sub-scales. the most pathological answer are rated 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, General Director, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided